CLINICAL TRIAL: NCT06041503
Title: A Phase II Multicenter Study of Enfortumab Vedotin With or Without Pembrolizumab in Rare Genitourinary Tumors (E-VIRTUE)
Brief Title: Enfortumab Vedotin With or Without Pembrolizumab in Rare Genitourinary Tumors (E-VIRTUE)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10001533; 001533-C
Record Dates: First submitted 2023-09-15; First posted 2023-09-18 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01-16

CONDITIONS: Adenocarcinoma of the Bladder; Squamous Cell Carcinoma of the Bladder; Testicular Germ Cell Tumors
Keywords: Immunotherapy; nectin 4; rare genitourinary cancers; programmed cell death 1 ligand 1
MeSH Terms: interventions — pembrolizumab; enfortumab vedotin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Treatment with enfortumab vedotin
  Interventions: Drug: Enfortumab vedotin
- Arm 2 (Experimental): Treatment with enfortumab vedotin and pembrolizumab
  Interventions: Drug: Pembrolizumab; Drug: Enfortumab vedotin

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is administered IV at 200 mg on day 1 of each 21-day cycle.
  Arms: Arm 2
Drug: Enfortumab vedotin — EV is administered IV at 1.25 mg/kg on days 1, 8, and 15 of each 28-day cycle (Arm 1) and on days 1 and 8 of each 21-day cycle (Arm 2).

SUMMARY:
Background:

Many cancers of the testicles and urinary tract are rare diseases; these are diseases that affect less than 200,000 people in the United States. It can be hard to study treatments for these diseases. One combination of drugs-enfortumab vedotin (EV) and pembrolizumab-has already been approved to treat some urinary cancers. Researchers want to see if they can help people with other types of testicle and urinary cancers.

Objective:

To test EV, with or without pembrolizumab, in patients with rarer cancers of the testicles or urinary tract.

Eligibility:

People aged 18 and older with rarer cancers of the testicles or urinary tract.

Design:

Participants will be screened. They will have a physical exam with blood and urine tests. Their ability to perform normal daily activities will be tested. They will have exams of their skin and eyes. They will have imaging scans. A biopsy may be needed: A sample of tissue will be removed from the tumor.

The study drugs are both given through a tube attached to a needle inserted into a vein in the arm. Some participants will receive treatments 3 times during 28-week cycles; others will receive treatments 2 times during 21-day cycles.

All participants may continue to receive treatments for up to 5 years. Imaging scans and other tests will be repeated.

Participants who stop taking the drugs will have follow-up visits every 3 to 4 weeks until the disease gets worse. They will have imaging scans and blood tests.

After that, follow-up visits will continue by phone every 3 months for up to 5 years after study therapy is finished.

DETAILED DESCRIPTION:
Background:

* Rare genitourinary (GU) tumors are tumors of aberrant histology occurring in the GU tract including kidney, bladder, ureters, testes, and penis. Due to their rarity, they are not systematically captured by currently available registries, treatment protocols or tissue banks.
* Large randomized clinical trials are logistically difficult in these small patient populations. Therefore, treatment information is obtained from case reports, retrospective studies, and small clinical trials, and is frequently extrapolated from trials on similar tumor types.
* Pembrolizumab is a potent and highly selective humanized monoclonal antibody that targets immune checkpoint programmed cell death protein 1 (PD-1) receptor.
* Nectin-4 is a type 1 transmembrane protein and member of a family of related immunoglobulinlike adhesion molecules implicated in cell-cell adhesion.
* Nectin-4 is highly expressed in cancer cells, particularly in urothelial carcinomas (UCs).
* Enfortumab vedotin (EV) is an antibody-drug conjugate consisting of a human monoclonal antibody to nectin-4 and monomethyl auristatin E (MMAE), a microtubule disrupting cytotoxic agent. EV has demonstrated a survival benefit in the setting of metastatic urothelial carcinoma, which has almost universally high nectin-4 expression.
* There is data in UC and bladder cancer variants showing co-existence of nectin-4 expression and programmed cell death 1 ligand 1 (PD-L1) expression and mismatch repair deficiency.
* There is currently very limited data on the level of nectin-4 expression in rare GU tumors and no evidence for the activity of EV in these tumors.

Objective:

-To assess the objective response rate (ORR) per RECIST v 1.1 in participants with rare genitourinary (GU) tumors treated with enfortumab vedotin (EV) with or without pembrolizumab.

Eligibility:

* Age >= 18 years
* Histologically confirmed diagnosis of locally advanced or metastatic pure adenocarcinoma of the urinary tract, pure squamous cell carcinoma of the urinary tract, or treatment-refractory testicular germ cell tumors.
* Participants may have received any number of prior anti-cancer treatments or be treatment na(SqrRoot) ve (with the exception of participants with testicular germ cell tumors, who must have exhausted all standard curative-intent options).

Design:

* This multisite study is a Phase II, open label, multicohort, nonrandomized study with two arms.
* Participants with:

  * Adenocarcinoma of the urinary tract will be enrolled in Cohort A (Cohort A1: prior anti-1/PD-L1 therapy; Cohort A2: no prior anti-PD-1/PD-L1 therapy).
  * Squamous cell carcinoma of the urinary tract will be enrolled in Cohort B (Cohort B1: prior anti-PD-1/PD-L1 therapy; Cohort B2: no prior anti-PD-1/PD-L1 therapy).
  * Testicular germ cell tumors will be enrolled in Cohort C (Cohort C1: prior anti-PD-1/PDL1 therapy; Cohort C2: no prior anti-PD-1/PD-L1 therapy).
* All participants will receive EV.
* Participants without prior immune checkpoint inhibitor (ICI) exposure will be eligible to receive concurrent pembrolizumab.
* Arm 1: EV monotherapy will be given in 28-day cycles for a maximum of 5 years, or until disease progression or intolerable side effects. EV will be administered I.V. at 1.25 mg/kg on days 1, 8, and 15 of each cycle.
* Arm 2: EV and pembrolizumab will be given in 21-day cycles. EV will be administered I.V. at 1.25 mg/kg on days 1 and 8 of each cycle. Pembrolizumab will be administered I.V. at 200 mg on day 1.

  * EV and pembrolizumab will be given for 35 cycles, or until a confirmed complete response, disease progression or intolerable side effects.
  * After the 35th cycle, EV may be continued to be given for a maximum of 5 years, or until disease progression or intolerable side effects.
  * Participants who have completed 35 cycles of pembrolizumab or stopped pembrolizumab for confirmed complete response may be eligible for up to additional 17 cycles of pembrolizumab if there is investigator-determined progressive disease by RECIST 1.1 after initial treatment.
* The accrual ceiling will be set at 68 participants to allow for inevaluable participants.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have histologically confirmed locally advanced or metastatic pure adenocarcinoma of the urinary tract, pure squamous cell carcinoma of the urinary tract, or treatment-refractory testicular germ cell tumors. Note: For the purposes of enrollment, the urinary tract is defined as the renal pelvis, ureter, bladder, and urethra.
* Participants must have measurable disease, per RECIST 1.1.
* Participants must have locally advanced or metastatic disease defined as new or progressive lesions on cross sectional imaging.
* Participants in Cohorts A1, B1, and C1 must have received prior anti-PD-1/PD-L1 therapy in any setting.
* Participants in Cohorts A2, B2, and C2 must be immune checkpoint inhibitor naive.
* Participants may be systemic treatment naive except for participants with testicular germ cell tumors, who must have received and be refractory to all standard options of curative-intent treatment.
* Age >= 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status <= 1 (Karnofsky >= 70%)
* Participants must have adequate organ and marrow function as defined below:

  * Hemoglobin (Hgb) >= 9g/dL
  * Absolute neutrophil count (ANC) >= 1,500/mcL
  * Platelets >= 100,000/mcL
  * Total bilirubin <= 1.5 x upper limit of normal (ULN) (<= 3 x ULN in participants with known/suspected Gilbert's disease)
  * Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) <= 2.5 x institutional ULN
  * Creatinine clearance (CrCl) >= 30 mL/min/1.73m^2 as estimated per institution standards.
* Pre-study treatment tissue availability (sufficient tissue for 25 unstained slides) is mandatory for enrollment. If tissue is determined to be insufficient/unsuitable, a fresh biopsy prior to study therapy will be required.
* Human immunodeficiency virus (HIV) positive participants are eligible if on stable dose of highly active antiretroviral therapy (HAART) for at least 3 months, CD4 counts are > 200 cells/mm^3 and viral load (VL) is undetectable.
* Hepatitis B virus (HBV) positive participants are eligible if they have been treated or are on an appropriate course of antivirals at study entry and with planned monitoring and management according to appropriate guidance. For previously treated participants or those with prior infection that has been cleared, prophylaxis is permitted, and hepatology consultation recommended.
* Hepatitis C virus (HCV) positive participants are eligible if participants are on active HCV therapy at study entry and on a stable dose of antivirals without documented clinically significant impaired liver function test or hematologic abnormalities and with planned monitoring and management according to appropriate labeling, or if they are post-treatment for HCV. Participants that are positive for hepatitis C must have a negative polymerase chain reaction (PCR).
* Women of child-bearing potential (WOCBP) must agree to use an effective method of contraception (barrier, surgical sterilization, abstinence prior to study entry, for the duration of study participation, and for at least 4 months after the last dose of study drug(s).
* Men able to father children must agree to use an effective method of contraception (barrier, surgical sterilization, abstinence) for the duration of the study treatment and up to 4 months after the last dose of the study drug(s). We also will recommend men with female partners of childbearing potential to ask female partners to be on an effective birth control (hormonal, intrauterine device (IUD), surgical sterilization).
* Breastfeeding participants must be willing to discontinue breastfeeding from study treatment initiation through 4 months after the last dose of the pembrolizumab and 3 weeks after the last dose of EV.
* Participants must be able to understand and willing to sign a written informed consent document.

EXCLUSION CRITERIA:

* Participants with prior investigational drug, chemotherapy, immunotherapy, or any prior radiotherapy (except for palliative bone directed therapy) within the past 2 weeks prior to the first study drug administration. Note: FDA-approved hormonal therapy for the treatment or prevention of other malignancies (e.g., breast cancer, prostate cancer) are allowed to be continued where in the opinion of the investigator stopping such therapies may increase the risk of disease progression. Potential drug-drug interactions with the hormonal agent will be assessed by the investigator prior to enrollment.
* Participants with prior treatment with EV or other MMAE-based ADCs.
* Participants with preexisting sensory or motor neuropathy Grade >= 2.
* History of severe allergic reactions attributed to compounds of similar chemical or biologic composition to EV and/or pembrolizumab.
* Symptomatic or untreated central nervous system (CNS) metastases. Note: Participants with previously treated brain or CNS metastases are eligible if the participants have recovered from any acute effects of radiotherapy and not requiring steroids, and any whole brain radiation therapy or any stereotactic radiosurgery was completed at least 2 weeks prior to initiation of study therapy.
* Participants will be excluded if they have an active autoimmune disease that might deteriorate when receiving pembrolizumab except for:

  * Diabetes type I, eczema, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment.
  * Participants requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses <= 10 mg of prednisone or equivalent per day.
  * Administration of steroids for other conditions through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation).
  * Participants on systemic intravenous or oral corticosteroid therapy with the exception of physiologic doses of corticosteroids (<= the equivalent of prednisone 10 mg/day) or other immunosuppressive agents such as azathioprine or cyclosporin A are excluded on the basis of potential immune suppression. For these participants these excluded treatments must be discontinued at least 1 week prior to treatment initiation for recent short course use (<= 14 days) or discontinued at least 4 weeks prior to treatment initiation for long term use (> 14 days). In addition, the use of corticosteroids as premedication for contrast-enhanced studies is allowed prior to treatment initiation and on study.
* History of uncontrolled diabetes mellitus within 3 months before the first dose of EV. Uncontrolled diabetes is defined as hemoglobin A1C (HbA1c) >= 8% or HbA1c between 7 and < 8% with associated diabetes symptoms (polyuria or polydipsia) that are not otherwise explained.
* Active keratitis or corneal ulcerations.
* Participants who have received or will receive a live vaccine within 30 days prior to the first administration of study intervention. Seasonal flu vaccines that do not contain a live virus are permitted. Locally approved COVID-19 vaccines are permitted.
* Pregnant women as evaluated by a positive serum or urine beta-human chorionic gonadotropin (Beta-hCG) test at screening.
* Participants with severe uncontrolled intercurrent illness that would limit compliance with study requirements, as evaluated by history, physical exam, and chemistry panel.
* Participants with severe uncontrolled intercurrent illness that would limit compliance with study requirements, as evaluated by history, physical exam, and chemistry panel. Participants with a prior (within 2 years of study therapy initiation) or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen will be permitted to join the study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | At every restaging (prior to every 2nd or 3rd cycle) until the end of the study therapy and during follow-up until PD
  Percentage of participants by best overall response (e.g., CR, PR, SD, PD) to therapy

SECONDARY OUTCOMES:
Second Objective response rate (ORR2) and second progression-free survival (PFS2) after second course of pembrolizumab | At every restaging (prior to every 2nd or 3rd cycle) until the end of the study therapy and during follow-up until PD
  Percentage of participants with the best overall response of CR or PR to therapy and duration of time from start of treatment to time of progression or death, whichever occurs first.
Duration of response (DoR) | At every restaging (prior to every 2nd or 3rd cycle) until the end of the study therapy and during follow-up until PD
  Time from start of treatment to disease progression or death in participants who achieve CR or PR
Overall survival (OS) | Day 1 of each cycle, at EoT, at the Safety visits, and every 90 days for up to a total of 5 years after the end of therapy.
  Time from the start of treatment that participants are still alive.
Progression-free survival (PFS) | At every restaging (prior to every 2nd or 3rd cycle) until the end of the study therapy and during follow-up until PD
  Duration of time from start of treatment to time of progression or death, whichever occurs first
Clinical benefit rate (CBR) | At every restaging (prior to every 2nd or 3rd cycle) until the end of the study therapy and during follow-up until PD
  Percentage of participant who have achieved CR, PR, and SD while on treatment.
Safety of EV with or without pembrolizumab | From first dose through 30 days after last treatment with EV and 90 days after last treatment with pembrolizumab
  Adverse events (AEs) will be reported by type and grade of toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Andrea B Apolo, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers at least 1 year after the completion of the primary endpoint.
Access Criteria: Data from this study may be requested by contacting the PI.

REFERENCES:
- [Derived] Chandran EBA, Atiq S, Simon N, Girardi D, Ley L, Cordes L, Patel R, Wang TF, Kydd AR, Redd B, Boudjadi S, Stukes I, Banday R, Smith E, Akbulut D, Niglio S, Gurram S, Steinberg S, Apolo AB. E-VIRTUE: a study of enfortumab vedotin with or without pembrolizumab in rare genitourinary tumors-design and rationale. Future Oncol. 2025 Jun;21(13):1625-1630. doi: 10.1080/14796694.2025.2497719. Epub 2025 May 27. PMID 40421891
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001533-C.html